CLINICAL TRIAL: NCT01651702
Title: Comparative Study of Two 3D Electroanatomical Mapping Systems for Ablations of Different Complex Arrhythmias
Brief Title: Comparison of Carto Versus Ensite 3D Electroanatomical Mapping Systems for Arrhythmias Ablations
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: Poor recruit rate
Sponsor: Rabin Medical Center (Other)
Responsible Party: Principal Investigator, Gregory Golovchiner, MD, Principle Invistigator, Rabin Medical Center
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0067-12-RMC
Record Dates: First submitted 2012-07-23; First posted 2012-07-27 (Estimated); Last update posted 2017-04-13 (Actual); Status verified 2017-04

CONDITIONS: Arrhythmias
Keywords: Arrhythmia; Electroanatomical mapping
MeSH Terms: conditions — Arrhythmias, Cardiac

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Carto (Active Comparator): Patients in whom Carto system will be used
  Interventions: Device: Carto
- Ensite (Active Comparator): Patients in whom Ensite system will be used
  Interventions: Device: Ensite

INTERVENTIONS:
Device: Carto — Group of patients where Carto Express system will be used for electroanatomical mapping.
  Arms: Carto
Device: Ensite — Group of patients where Ensite Velocity system will be used for electroanatomical mapping.
  Arms: Ensite

SUMMARY:
Three dimensional anatomical mapping is an established method facilitating ablation of cardiac arrhythmias. The most commonly used systems are CARTO® System (Biosense Webster, Inc., Diamond Bar, CA, USA) and EnSite NavX™ (St. Jude Medical, Inc., St. Paul, MN, USA). These two systems has been compared in only a few studies. Recent technical advances resulted in the development of new versions of both systems. To the best of the investigators knowledge no studies have been performed for direct comparison of the newer versions of these two systems. The aim of the study to compare two systems for the use in the ablation of complex arrhythmias.

DETAILED DESCRIPTION:
Background:

Three dimensional anatomical mapping is an established method facilitating ablation of cardiac arrhythmias. It is nowadays an excepted method especially for complex arrhythmias such as atrial fibrillation and ventricular tachycardia.

The most commonly used systems are CARTO® System (Biosense Webster, Inc., Diamond Bar, CA, USA) and EnSite NavX™ (St. Jude Medical, Inc., St. Paul, MN, USA). These mapping systems have helped to decrease procedural complexity, procedure time, and improve safety. The EnSite NavX system uses impedance measurements between the individual catheter electrodes and the patches placed on the patient's chest and abdomen. The CARTO system utilizes magnetic location technology to provide accurate visualization of the magnet sensor-equipped catheter tip.

These two systems has been compared in only a few studies. Different results have been found in simple ablations versus more complex ablation of atrial fibrillation. Recent technical advances resulted in the development of new versions of both systems. Carto Express version allows quicker mapping and reconstruction of heart cavities and great vessels geometry as compared to previous versions of Carto XP. EnSite Velocity system incorporates more precise catheter visualization, and allows quicker mapping as compared to previous version of EnSite.

To the best of the investigators knowledge no studies have been performed for direct comparison of the newer versions of these two systems.

Study design Prospective single-center non-randomized open label comparison study. Primary objective Comparison of Carto Express system vs. EnSite Velocity system for ablation of complex arrhythmias.

End points:

1. Procedure duration.
2. Fluoroscopy time
3. Procedure success -will be measured in terms of the 1-year recurrent arrhythmia rate Study population Patients planned for ablation of complex arrhythmia.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18- 80.
2. Ability to sign informed consent.
3. History of one of the following arrhythmias requiring the use of 3D electroanatomical mapping:

   * Symptomatic paroxysmal or persistent atrial fibrillation with failed treatment of at least two anti-arrhythmic drugs.
   * Ischemic ventricular tachycardia necessitating ablation as per decision of electrophysiologist.
   * Symptomatic atrial tachycardia after failed medical treatment.
   * Symptomatic idiopathic ventricular tachycardia.

Exclusion Criteria:

1. Unstable patients not allowing performing procedure more than 2 hours
2. Patients planned for one of the two systems compared for whatever reason Ex. procedure planned with NAVX system Array Balloon).

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2015-07; Primary Completion 2016-07 (Estimated); Study Completion 2016-10 (Estimated)

PRIMARY OUTCOMES:
Procedure duration | Procedure duration - average expected 2.5 hours
  Average procedure duration (needle to catheters withdrawal)

SECONDARY OUTCOMES:
Fluoroscopy time | Procedures will be evaluated for the fluoro time, expected average 30 min
  Average fluro time in each of groups.
Procedure success | Patients will be followed for one year for recurrency of arrhythmia
  Recurrency of the arrhythmia assessed by blinded electrophysiologist

CONTACTS AND LOCATIONS:
Overall Officials: Gregory Golovchiner, MD, Principal Investigator — Rabin Medical Center